CLINICAL TRIAL: NCT00512018
Title: Neuromuscular Electrical Stimulation and Isokinetic Training: Effects on Strength and Neuromuscular Properties
Brief Title: Neuromuscular Electrical Stimulation and Isokinetic Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Mariana Arias Avila, MSc, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 067/03
Record Dates: First submitted 2007-08-03; First posted 2007-08-07 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
Keywords: Electric Stimulation; Quadriceps Muscle; Muscle Strength; Neuromuscular Properties; Tension-Length Relationship; Healthy young adults

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isokinetic Exercise only (Active Comparator): Individuals were asked to perform a 8-session training, twice a week, in which they trained the knee extensors muscles in an isokinetic dynamometer, 3 sets of 10 repetitions.
  Interventions: Other: Isokinetic exercise
- Isokinetic exercise + NMES (Experimental): In the contralateral limb, the same protocol was repeated; however, each contraction was associated with overlapped NMES (Ex+NMES).
  Interventions: Device: NMES

INTERVENTIONS:
Device: NMES — In the contralateral limb, the same protocol was repeated; however, each contraction was associated with overlapped NMES (Ex+NMES limbs).For the NMES, a symmetric double-phase sine-wave was used. Bearing wave frequency was of 2500 Hz, modulated in 50 bursts/s, with pulse duration of 200 µs, interburst interval of 10 ms. This configuration is known as "Russian current".
  Other Names: Current generator Physiotonus Slim (Bioset, Brazil)
  Arms: Isokinetic exercise + NMES
Other: Isokinetic exercise — Subjects realized training sessions twice a week with a 2-day minimum interval between the sessions, for 4 weeks. Each session included 5 min period of warm-up in a stationary bicycle, followed by 3 series of quadriceps stretching, as previously described. After being positioned at the isokinetic dynamometer, just as in the evaluation sessions, subjects firstly performed 3 sets of 10 maximum isokinetic concentric repetitions at the speed of 30º/s with one limb (EX limb), respecting the rest interval of 3 minutes between the sets.
  Other Names: Isokinetic Dynamometer: Biodex Multi Joint System 3
  Arms: Isokinetic Exercise only

SUMMARY:
The purpose of this study was to assess the effects of Neuromuscular Electrical Stimulation (NMES) associated to an isokinetic training program in both young healthy men and women. Twenty subjects (10 men, 10 women; 21±1.5 years) submitted both quadriceps femoris muscles to a strengthening program (3 sets of 10 isokinetic concentric repetitions at 30°/s) two days per week for 4 weeks. One limb was submitted only to the strength training (EX) while the other underwent the same training program but with NMES added to each contraction (Ex+NMES). The current used for NMES was Russian Current (frequency of 2500 Hz, 50 bursts/s and pulse duration of 200 µs). The evaluation protocol included isometric and isokinetic concentric extensor torques at 30°/s. Men increased their torque in both tested modalities in both limbs, with no difference between them. The angle of peak torque increased for the EX limb, showing an altered tension-length relationship, which did not occur for the Ex+NMES limb or for women. Women increased their torque for EX limb in both modalities, which only occured for isometric mode in the Ex+NMES limb. However, they showed a decrease in their acceleration time in Ex+NMES limbs, showing they could produce a muscular contraction more readily than they did before training. The results of this study found that the association between NMES and isokinetic concentric voluntary strength training does not improve strength gains of voluntary training itself for young healthy subjects of both genders. However, it could improve neuromuscular readiness to produce torque in women.

DETAILED DESCRIPTION:
Subjects Twenty active and healthy undergraduate students (men: 21 ± 1.9 years; 1.77 ± 0.1 m; 73 ± 8.4 kg; 23.3 ± 1.4 kg/m²; women: 20.9 ± 0.7 years; 1.64 ± 0.1 m; 56.3 ± 5.5 kg; 21 ± 1.0 kg/m²) were selected for this study. All of them underwent physical examination before the study and had already participated in strength training programs before this study. All 10 men selected concluded the study. Although 15 women were selected and began the training program, 5 were excluded: 3 reported episodes of pain in the knee joint during training sessions, and 2 of them could not conclude the training program for personal reasons. Therefore, the final data refers to 10 women.

All procedures for evaluation and training were explained before and a consent term was signed. The project was approved by the Ethics Committee for Medical Research of Federal University of São Carlos and is in agreement with the Declaration of Helsinki.

Evaluation protocol Before all evaluations, subjects were familiarized with testing and training procedures. All the evaluation and training procedures were applied for both right and left limbs of subjects before and after training program. To avoid possible dominance effects, volunteers were randomly separated to determine in which limb (right or left) training would be associated with NMES. The investigator who made the data analysis was blind to this randomization.

After 5 min period of warm-up in a stationary bicycle at a speed of 20 km/h and load of 20 W, the subjects stretched the quadriceps femoris and the hamstring muscles of both limbs. Each muscle group was stretched 3 times of 30 s alternately. Afterwards, the subject was positioned in an isokinetic dynamometer (Biodex® Multi-joint System 3, Biodex, Shirley, NY), with the angulation of 100º on hips. Trunk, pelvis, and thigh of subjects were stabilized by strips, following equipment description36. Rotation axis of dynamometer was aligned with axis of the knee, at the level of lateral epicondyle of the femur, while the attachment was fixed at the distal part of leg of subjects, about 5 cm above medial malleolus. The gravity effect correction was calculated with the limb at 60° of flexion. The isokinetic device was calibrated before each evaluation and training session as requested by the manufacturer.

After that, volunteers had their knees positioned at 60° and were familiarized to the action they would do. After that, they were asked to perform 3 maximum voluntary isometric knee extension contractions for 5 s, with 1 min of rest interval between the contractions. Three min after the last contraction, subjects were familiarized with the isokinetic contraction and then performed 5 maximum isokinetic concentric knee extension contractions at 30º/s speed, from 90° to 15°, 0° being full extension, totaling up 75° of Range of Motion (ROM). Verbal encouragement37 as well as visual feedback from the equipment38 were given in an attempt to achieve a maximal voluntary effort level during all contractions each subject was asked to perform. The same procedures were repeated with the contralateral limb.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were to be young (age range between 18 and 25 years), body mass index considered normal (between 20 and 25 kg/m²), practice of physical activity other than resistance training during the training period, absence of any neuromuscular disorders in lower limbs, no knee pain history.

Exclusion Criteria:

* The exclusion criteria were pregnancy, epilepsy, cancer, and suspicion on heart disease, recent surgery, respiratory disorders, non-compensated diabetes, and history of trauma, fracture or surgery in lower limbs, reports of pain at knee joint.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2005-01; Primary Completion 2006-12 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The association between NMES and isokinetic concentric voluntary strength training did not improve strength gains of voluntary training itself for young healthy subjects of both genders. | Six months after stopping other type of strength training

CONTACTS AND LOCATIONS:
Overall Officials: Mariana A Avila, PT, Principal Investigator — Universidade Federal de Sao Carlos; Tania F Salvini, PhD, Study Director — Universidade Federal de Sao Carlos; Jamilson S Brasileiro, PhD, Study Chair — Universidade Federal do Rio Grande do Norte